CLINICAL TRIAL: NCT03631082
Title: Effects of Slump Stretching vs Lumbar Mobilization With Exercises in Relieving Non-radiculating Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Isra University (Other)
Responsible Party: Principal Investigator, Sundus Iftikhar, Research Associate, Isra University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIRS-IUISB/SMMPT/001
Record Dates: First submitted 2018-08-12; First posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Low Back Pain
Keywords: effects; slump stretching; lumbar mobilization; non radiculating; Low back pain; exercises; quality of life; modified oswestry low back pain disability; numeric pain rating scale; fear avoidance beliefs
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: The two groups will be Slump stretching group and Lumbar mobilization group. All physical therapy techniques in both groups will be applied 3 times in a week up to 2 weeks with each session consisting of 25-40 minutes.
  Group 1 will receive slump stretching along with standardized exercises while group 2 will recieve lumbar mobilization along with standardized exercises.
  Demographic details of the patients will be collected at baseline (1st Visit) while Modified Oswestry Low Back Pain Disability Questionnaire,Numeric pain rating scale,Fear-Avoidance Beliefs Questionnaire,Active range of motion (AROM) of lumbar spine and Short-Form Health Survey (SF-36) will be measured at baseline, 1st week, and final week.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Slump stretching group (Experimental): Slump stretching will be performed with the patient in the long sitting position. The position will be held for 30 seconds. A total of 5 repetitions will be completed.
  Patients will also complete a standardized exercise program consisting of pelvic tilts, bridging, wall squats, and quadruped alternate arms/legs activities as described by Cleland et al.
  Patients will perform 10 repetitions of each exercise.
  Interventions: Other: Slump stretching
- Lumbar mobilization group (Active Comparator): Maitland Grade 1 - 2 Posterior to anterior lumbar spine mobilization will be applied for 30 - 45 seconds for all segments through L1 to L5 at rate of 1 oscillation per 2 seconds.
  Patients will also complete a standardized exercise program consisting of pelvic tilts, bridging, wall squats, quadruped alternate arms/legs activities as described by Cleland et al.
  Patients will perform 10 repetitions of each exercise.
  Interventions: Other: Lumbar mobilization

INTERVENTIONS:
Other: Slump stretching — Slump stretching will be provided to this group along with standardized exercises.
  Arms: Slump stretching group
Other: Lumbar mobilization — Lumbar mobilizations will be provided to this group along with standardized exercises.
  Arms: Lumbar mobilization group

SUMMARY:
This study will be conducted to determine the effects of slump stretching vs lumbar mobilization with exercises in relieving non-radiculating low back pain. There will be two groups; Group I will receive Slump stretching along with standardized exercises and Group II will receive Lumbar mobilizations along with standardized exercises.

DETAILED DESCRIPTION:
Physical therapist commonly examines and treats patients with low back pain. For this purpose, they utilize a wide range of interventions for the management of Low back pain.

The rhythmical movement is thought to modulate pain and muscle spasm by stimulating receptors within the mobilized structures while, In recent years, neurodynamic test procedures, have also been used as interventions to potentially resolve abnormal physiology within the nervous system.

So for this purpose not only the present study can provide an additional evidence to the literature but also can can also demonstrates a structured Physiotherapy plan for treating the Non-Radiculating Low back pain

ELIGIBILITY:
Inclusion Criteria:

Individuals with Non-Radiculating Low back pain

Test:

i. Slump test=positive ii. Straight leg raise=negative

Exclusion Criteria:

Individuals with Radiculating Low Back pain,History of spinal surgery, Disc herniation,Pregnant women, Major diseases (e.g. stroke)

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Numeric pain rating scale | 2 weeks
  On a scale of 0 to 10, with 0 being no pain at all and 10 being the worst pain imaginable.
Modified Oswestry Low Back Pain Disability Questionnaire | 2 weeks
  The questionnaire has been designed to give the therapist information as to how the back pain has affected the ability to manage in everyday life.
Short-Form Health Survey (SF-36) | 2 weeks
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting.

SECONDARY OUTCOMES:
Fear-Avoidance Beliefs Questionnaire | 2 weeks
  It consist of two scales; Scale 1: fear-avoidance beliefs about work Scale 2: fear-avoidance beliefs about physical activity
Active range of motion of lumbar spine. | 2 weeks
  It includes; lumbar flexion lumbar extension left lateral flexion right lateral flexion

IPD SHARING:
Plan to Share IPD: Undecided